CLINICAL TRIAL: NCT02553941
Title: Phase 1b Trial of the Combination of Ibrutinib and Azacitidine for the Treatment of Higher Risk Myelodysplastic Syndromes in Previously Treated Patients or in Untreated Patients Unfit for or Who Refuse Intense Therapy
Brief Title: Ibrutinib and Azacitidine for Treatment of Higher Risk Myelodysplastic Syndrome
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Brian Jonas (Other)
Collaborators: Pharmacyclics LLC. (Industry)
Responsible Party: Sponsor-Investigator, Brian Jonas, Principal Investigator, University of California, Davis
Organization: University of California, Davis (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 755461; UCDCC#256 (Other: UC Davis); PCI-32765 (Other: UCDCC); UCDCC#256 (Other: University of California Davis Comprehensive Cancer Center)
Record Dates: First submitted 2015-07-27; First posted 2015-09-18 (Estimated); Last update posted 2022-10-06 (Actual); Status verified 2022-10

CONDITIONS: Chronic Myelomonocytic Leukemia; de Novo Myelodysplastic Syndrome; Previously Treated Myelodysplastic Syndrome; Refractory Anemia With Excess Blasts in Transformation; Secondary Myelodysplastic Syndrome
MeSH Terms: conditions — Leukemia, Myelomonocytic, Chronic | interventions — Azacitidine; ibrutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- azacitidine, ibrutinib (Experimental): Patients receive azacitidine intravenous infusion over 10-40 minutes or subcutaneous on days 1-7 or 1-5 and 8-9, and ibrutinib by mouth one daily on days 1-28. Treatment repeats every 28 days for up to 24 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Azacitidine; Drug: Ibrutinib

INTERVENTIONS:
Drug: Azacitidine — Given intravenous or subcutaneous
  Other Names: Vidaza
Drug: Ibrutinib — Given by mouth once daily
  Other Names: BTK Inhibitor

SUMMARY:
This phase Ib trial studies the side effects and best dose of ibrutinib when given together with azacitidine in treating patients with myelodysplastic syndrome that is likely to occur or spread (higher risk) and who were previously treated or untreated and unfit for or refused intense therapy. Ibrutinib and azacitidine may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the safety and tolerability of ibrutinib in combination with azacitidine in patients with higher risk myelodysplastic syndrome (MDS) and to determine the maximum tolerated dose (MTD) or recommended Phase 2 dose of ibrutinib combined with azacitidine.

SECONDARY OBJECTIVES:

I. To do an early assessment of the efficacy of the combination of ibrutinib and azacitidine in higher risk MDS. Specific secondary endpoints include: disease response per modified International Working Group (IWG) 2006 response criteria for MDS, hematologic normalization rate (HNR = complete remission [CR] + partial remission [PR] + hematologic improvement [HI]), overall survival (OS), progression free survival (PFS), disease free survival (DFS), and time to response (TTR).

TERTIARY OBJECTIVES:

I. To evaluate the pharmacodynamic and biological effects and impact of quality of life (QoL) of the combination of ibrutinib and azacitidine in patients with higher risk MDS is the exploratory objective of this study. Exploratory endpoints include: laboratory biomarker analysis and effect on QoL assessments.

OUTLINE: This is a dose-escalation study of ibrutinib.

Patients receive azacitidine intravenously (IV) over 10-40 minutes or subcutaneously (SC) once daily (QD) on days 1-7 or 1-5 and 8-9, and ibrutinib orally (PO) QD on days 1-28. Treatment repeats every 28 days for up to 24 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months for 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed diagnosis of myelodysplastic syndrome
* Revised international prognostic scoring system (IPSS-R) intermediate, high or very high
* For the dose escalation cohorts, any prior number of MDS therapies, including hypomethylating agents, are permitted; for the dose expansion cohort, subjects must be azacitidine naïve, but otherwise any prior number of MDS therapies are permitted; treatment naïve patients are eligible for both the dose escalation and expansion cohorts if they are unfit for or refuse intense therapy
* No specific hematologic parameters for study entry are required; transfusion-dependent patients are eligible and platelet counts should be maintained greater than 10,000/mm^3
* Serum aspartate transaminase (AST) and alanine transaminase (ALT) =< 3.0 x upper limit of normal (ULN)
* Estimated creatinine clearance >= 30 ml/min (Cockcroft-Gault)
* Bilirubin =< 1.5 x ULN (unless bilirubin rise is due to Gilbert's syndrome or of non-hepatic origin)
* Prothrombin time (PT)/international normalized ratio (INR) < 1.5 x ULN and partial thromboplastin time (PTT) (activated [a]PTT) < 1.5 x ULN
* Karnofsky performance status (KPS) performance status of 60% or greater
* Female subjects who are of non-reproductive potential (ie, post-menopausal by history - no menses for >= 1 year; OR history of hysterectomy; OR history of bilateral tubal ligation; OR history of bilateral oophorectomy); or, female subjects of childbearing potential must have a negative serum pregnancy test upon study entry
* Male and female subjects who agree to use highly effective methods of birth control during the period of therapy and for 30 days after the last dose of study drug

Exclusion Criteria:

* Known bleeding disorders, active bleeding disorders or clinical signs of bleeding (grade >= 2)
* Prior bone marrow transplant within 3 months or with acute graft versus host disease (GVHD)
* Prior treatment with a Bruton's tyrosine kinase (BTK) inhibitor
* Anticancer therapy including chemotherapy, immunotherapy, radiotherapy, hormonal or any investigational therapy within 14 days or 5 half-lives prior to first dose of study drug
* Unresolved toxicities from prior anti-cancer therapy, defined as having not resolved to Common Terminology Criteria for Adverse Event (CTCAE, version 4.03), grade =< 1, or to the levels dictated in the inclusion/exclusion criteria with the exception of alopecia
* History of other malignancies, except:

  * Malignancy treated with curative intent and with no known active disease present for >= 1 years before the first dose of study drug and felt to be at low risk for recurrence by treating physician
  * Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease
  * Adequately treated carcinoma in situ without evidence of disease
  * Low-risk prostate cancer after curative surgery
* Concurrent systemic immunosuppressant therapy
* Vaccinated with live, attenuated vaccines within 4 weeks of first dose of study drug
* Recent infection requiring intravenous systemic treatment
* History of stroke or intracranial hemorrhage within 6 months prior to enrollment
* Known history of human immunodeficiency virus (HIV) or active with hepatitis C virus (HCV) or hepatitis B virus (HBV); subjects who are positive for hepatitis B core antibody or hepatitis B surface antigen must have a negative polymerase chain reaction (PCR) result before enrollment; those who are PCR positive will be excluded
* Major surgery within 4 weeks of first dose of study drug
* Any life-threatening illness, medical condition, or organ system dysfunction that, in the investigator's opinion, could compromise the subject's safety or put the study outcomes at undue risk
* Currently active, clinically significant cardiovascular disease, such as uncontrolled arrhythmia or class 3 or 4 congestive heart failure as defined by the New York Heart Association Functional Classification; or a history of myocardial infarction, unstable angina, or acute coronary syndrome within 6 months prior to enrollment
* Unable to swallow capsules or malabsorption syndrome, disease significantly affecting gastrointestinal function, or resection of the stomach or small bowel, symptomatic inflammatory bowel disease or ulcerative colitis, or partial or complete bowel obstruction
* Concomitant use of warfarin or other vitamin K antagonists
* Requires treatment with a strong cytochrome P450 (CYP) family 3, subfamily A, polypeptide 4/5 (3A4/5) inhibitor
* Lactating or pregnant
* Unwilling or unable to participate in all required study evaluations and procedures
* Unable to understand informed consent form (ICF)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2016-05-17 (Actual); Primary Completion 2019-05-25 (Actual); Study Completion 2019-11-07 (Actual)

PRIMARY OUTCOMES:
Incidence of toxicity of ibrutinib and azacitidine, graded according to the Common Terminology Criteria for Adverse Events | Within 30 days following the last dose of study drug or the first date starting new anticancer therapy
  For each adverse event, the percentage of subjects who experience at least 1 occurrence of the given event will be summarized.

SECONDARY OUTCOMES:
Disease Free Survival | From the time of first documented Complete Response until relapse or the date of death from any cause, assessed up to 6 months post-treatment
  For subjects achieving a Complete Response, Disease Free Survival will be calculated to determine durability of response. Descriptive statistics will be used, including mean, standard deviation, median, and minimum and maximum values for continuous variables and frequencies and percentages for categorical variables. Time-to-event data will be summarized descriptively by life-table statistics (median time to event; Kaplan-Meier plots).
Disease response per modified International Working Group (IWG) 2006 response criteria for MDS | Up to 96 weeks
  Descriptive statistics will be used, including mean, standard deviation, median, and minimum and maximum values for continuous variables and frequencies and percentages for categorical variables.
HNR, defined as the proportion of treated subjects who achieve a CR, PR or HI as best response as assessed by the investigator and as defined by the modified IWG 2006 response criteria for MDS | Up to 96 weeks
  Descriptive statistics will be used, including mean, standard deviation, median, and minimum and maximum values for continuous variables and frequencies and percentages for categorical variables.
Overall survival | From the time of first study drug administration until the date of death from any cause, assessed up to 6 months post-treatment
  Descriptive statistics will be used, including mean, standard deviation, median, and minimum and maximum values for continuous variables and frequencies and percentages for categorical variables. Time-to-event data will be summarized descriptively by life-table statistics (median time to event; Kaplan-Meier plots).
Progression Free Survival | From the time of first study drug administration until the date of progression or death from any cause, assessed up to 6 months post-treatment
  Descriptive statistics will be used, including mean, standard deviation, median, and minimum and maximum values for continuous variables and frequencies and percentages for categorical variables. Time-to-event data will be summarized descriptively by life-table statistics (median time to event; Kaplan-Meier plots).

OTHER OUTCOMES:
Change in biomarker levels including BTK, phosphatidylinositol 3 kinase, cluster of differentiation 34, mitogen-activated protein kinase, nuclear transcription factor kappa-B, interleukin 2-inducible T-cell kinase, and peripheral T cells and subsets | Baseline up to 96 weeks
  Laboratory tests will be summarized separately for hematology and serum chemistry. Descriptive statistics will be provided for the values of selected clinical laboratory tests at each scheduled on-treatment evaluation including the final value. Percent change from baseline to each scheduled on-treatment evaluation and to the final value will also be summarized. For selected variables, the mean value and mean percent change over time will be presented graphically. All laboratory values will be converted to standard international units and will be graded using the NCI CTCAE version 4.03.
Quality of LIfe of the combination of ibrutinib and azacitidine, assessed by the European Organization for Research and Treatment of Cancer Quality of Life Questionnaires | Up to 30 days from last dose

CONTACTS AND LOCATIONS:
Overall Officials: Brian Jonas, Principal Investigator — University of California, Davis
Locations (5):
- United States (5):
  - UCLA / Jonsson Comprehensive Cancer Center, Los Angeles, California
  - UC Irvine Health/Chao Family Comprehensive Cancer Center, Orange, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - University of California San Diego, San Diego, California
  - University of California, San Francisco, San Francisco, California